CLINICAL TRIAL: NCT01119716
Title: International Registry on Cardioversion of Atrial Fibrillation
Brief Title: International Registry on Cardioversion of Atrial Fibrillation (MK-6621-051)
Acronym: RHYTHM-AF
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Institut für Herzinfarktforschung an der Universität Heidelberg (Unknown)
Responsible Party: Sponsor
Other Study IDs: 6621-051; 2010_025
Record Dates: First submitted 2010-05-06; First posted 2010-05-07 (Estimated); Results first posted 2014-01-30 (Estimated); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; Afib; cardioversion; normal sinus rhythm; arrhythmia; AF
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Enrolled Participants: Participants with documented atrial fibrillation in the hospital setting for whom a cardioversion is one of the planned therapeutic options

SUMMARY:
This study will create a prospective registry of consecutive patients with Atrial Fibrillation (Afib) considered for cardioversion treatment to document up-to-date practice of in-hospital treatment, with a focus on the characterization of type of Afib, as well as on treatments applied (drugs, devices, interventions and their combinations), and associated complications within 60 days after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Participant with documented atrial fibrillation (confirmed by electrocardiogram) in the hospital setting at the time of enrollment
* Planned cardioversion (of atrial fibrillation)

Exclusion Criteria:

* Already enrolled in this or any other clinical trial
* Atrial flutter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in a hospital setting in Australia, Brazil, France, Germany, Italy, Netherlands, Poland, UK, Spain, and Sweden from a cross section of different centers including university and non-university hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 4658 (Actual)
Dates: Start 2010-05-25 (Actual); Primary Completion 2013-02-15 (Actual); Study Completion 2013-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Crijns HJ, Weijs B, Fairley AM, Lewalter T, Maggioni AP, Martin A, Ponikowski P, Rosenqvist M, Sanders P, Scanavacca M, Bash LD, Chazelle F, Bernhardt A, Gitt AK, Lip GY, Le Heuzey JY. Contemporary real life cardioversion of atrial fibrillation: Results from the multinational RHYTHM-AF study. Int J Cardiol. 2014 Apr 1;172(3):588-94. doi: 10.1016/j.ijcard.2014.01.099. Epub 2014 Jan 25. PMID 24556445
- [Derived] Crijns HJ, Bash LD, Chazelle F, Le Heuzey JY, Lewalter T, Lip GY, Maggioni AP, Martin A, Ponikowski P, Rosenqvist M, Sanders P, Scanavacca M, Bernhardt AA, Unniachan S, Phatak HM, Gitt AK. RHYTHM-AF: design of an international registry on cardioversion of atrial fibrillation and characteristics of participating centers. BMC Cardiovasc Disord. 2012 Oct 2;12:85. doi: 10.1186/1471-2261-12-85. PMID 23031215

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with documented atrial fibrillation in the hospital setting for whom a cardioversion is one of the planned therapeutic options
Period: Overall Study
Arm/Group | All Enrolled Participants
Started | 4658
Completed | 4658
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 4658
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1742
  Male | 2916

OUTCOME MEASURES:

1. Primary Outcome: Cardiovascular Disease History of Participants Presenting With Atrial Fibrillation at Baseline (Admission)
Time Frame: Baseline (time of admission)
Population: All enrolled participants with baseline cardiovascular history data.
Measure: Number; unit: Percentage of Participants
Groups:
- Male: Male participants with documented atrial fibrillation in the hospital setting for whom a cardioversion is one of the planned therapeutic options
- Female: Female participants with documented atrial fibrillation in the hospital setting for whom a cardioversion is one of the planned therapeutic options
- Total: All participants with documented atrial fibrillation in the hospital setting for whom a cardioversion is one of the planned therapeutic options
Arm/Group | Male | Female | Total
Number analyzed (Participants) | 2909 | 1740 | 4649
Percentage of Participants
  Congenital Heart Disease | 1.3 | 1.6 | 1.4
  Sick Sinus Syndrome | 2.3 | 3.5 | 2.8
  Sustained Ventricular Tachycardia | 1.2 | 0.5 | 0.9
  Ventricular Fibrillation | 0.7 | 0.4 | 0.6

2. Primary Outcome: Co-Morbidity in Participants Presenting With Atrial Fibrillation at Baseline (Admission)
Time Frame: Baseline (time of admission)
Population: All enrolled participants with co-morbity data available.
Measure: Number; unit: Percentage of Participants
Arm/Group | Male | Female | Total
Number analyzed (Participants) | 2851 | 1711 | 4562
Percentage of Participants
  Chronic Obstructive Pulmonary Disease | 7.8 | 7.1 | 7.5
  Peripheral Vascular Disease | 6.3 | 5.1 | 5.8
  Chronic Renal Failure | 6.7 | 5.3 | 6.2
  Anemia | 3.6 | 5.3 | 4.2
  Sleep Apnea Syndrome | 4.8 | 2.1 | 3.8
  Haemorrhagic Complication | 1.2 | 1.8 | 1.4

3. Primary Outcome: Clinical Type of Atrial Fibrillation at Baseline (Admission)
Time Frame: Baseline (time of admission)
Population: All enrolled participants with admission (baseline) atrial fibrillation data available.
Measure: Number; unit: Percentage of Participants
Arm/Group | Male | Female | Total
Number analyzed (Participants) | 2909 | 1740 | 4649
Percentage of Participants
  1st Detected Episode | 29.2 | 33.6 | 30.8
  Paroxysmal | 27.2 | 31.9 | 28.9
  Persistent | 36.4 | 27.6 | 33.1
  Permanent | 4.2 | 3.6 | 4.0
  Unknown | 3.0 | 3.3 | 3.1

4. Primary Outcome: Treatments Utilized for Participants for Atrial Fibrillation
Time Frame: At time of Treatment (up to 1 day from admission)
Population: All enrolled participants with available data pertaining to type of therapy(s) used to treat the participants atrial fibrillation.
Measure: Number; unit: Participants
Arm/Group | Male | Female | Total
Number analyzed (Participants) | 2916 | 1742 | 4658
Participants
  Electrical Cardioversion | 1677 | 792 | 2469
  Pharmacological Cardioversion | 705 | 609 | 1314
  Combined Electrical/Pharmacological Cardioversion | 120 | 69 | 189
  Rate Control Change | 215 | 152 | 367
  Catheter Ablation | 92 | 32 | 124
  Surgical Therapy | 1 | 0 | 1
  Implantable Cardiac Defibrillator | 10 | 0 | 10
  Pacemaker | 20 | 18 | 38
  No Treatment | 550 | 342 | 892

5. Primary Outcome: Percentage of Participants Who Had a Successful Electrical or Pharmacological Cardioversion
Description: Pharmacological cardioversion was considered successful if sinus rhythm or atrial rhythm was obtained within 24 hours after its initiation. Electrical cardioversion was considered successful if sinus rhythm was obtained and maintained for at least 10 minutes after the last shock was administered.
Time Frame: At time of treatment (up to 1 day from admission)
Population: Participants who had artrial fibrillation treated by either electrical or pharmacological cardioversion.
Measure: Number; unit: Percentage of Participants
Groups:
- Male: Male participants with documented atrial fibrillation in the hospital setting for whom an electrical or pharmacological cardioversion was perfomed
- Female: Female participants with documented atrial fibrillation in the hospital setting for whom an electrical or pharmacological cardioversion was perfomed
Arm/Group | Male | Female | Total
Number analyzed (Participants) | 2262 | 1332 | 3594
Percentage of Participants
  Electrical Cardioversion | 69.5 | 55.1 | 64.2
  Pharmacological Cardioversion | 30.5 | 44.9 | 35.8

6. Primary Outcome: Complications Experienced by Participants Who Underwent a Cardioversion for Treatment of Atrial Fibrillation
Time Frame: up to 60 days from day of treatment (cardioversion)
Population: All enrolled participants with follow-up data available
Measure: Number; unit: Participants
Arm/Group | Male | Female | Total
Number analyzed (Participants) | 2633 | 1507 | 4140
Participants
  Myocardial Infarction | 2 | 2 | 4
  Non-haemorrhagic Stroke | 7 | 3 | 10
  Haemorrhagic Stroke | 1 | 0 | 1
  Peripheral Embolism | 0 | 2 | 2
  Pulmonary Embolism | 1 | 3 | 4
  Transient Ischaemic Attack | 0 | 1 | 1
  Heart Failure | 9 | 10 | 19
  Major Bleeding | 3 | 3 | 6
  Minor Bleeding | 12 | 6 | 18
  Recurrence of Atrial Fibrillation | 107 | 63 | 170
  Recurrence of Atrial Flutter | 10 | 2 | 12
  Asystole for more than 3 seconds | 2 | 2 | 4
  Symptomatic Ventricular Tachycardia | 0 | 1 | 1
  Ventricular Fibrillation | 2 | 1 | 3
  Sick Sinus syndrome | 1 | 2 | 3
  Torsade de pointes | 0 | 1 | 1
  Syncope | 5 | 4 | 9
  Endocarditis | 0 | 1 | 1
  Tamponade | 1 | 0 | 1
  Bradycardia | 4 | 0 | 4
  Hypotension | 4 | 1 | 5
  Other Complication | 27 | 18 | 45
  Death | 198 | 113 | 311

ADVERSE EVENTS:
Description: No formal reporting or recording of adverse events was conducted during this observational study.
Arm/Group | All Enrolled Participants
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Scientific Committee for the study has the authority to make all decisions related to design, conduct, data interpretation and dissemination of study results.